CLINICAL TRIAL: NCT06809738
Title: Proposal for an Anatomical Scale for the Prognosis of Fournier Syndrome.
Brief Title: Anatomical Scale for the Prognosis of Fournier Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Huber Díaz Fuentes, Urologist, Instituto Mexicano del Seguro Social
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2311
Record Dates: First submitted 2025-01-26; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Fournier's Gangrene
Keywords: Surgery; Infection; tissue; scrotal
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: 3-stage reconstructive technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: reconstructive technique — 1. Analysis and limitation of the tissue injury. Bilateral testicular and spermatic cord dissection.
  2. Formation of cutaneous flaps and bilateral inguinal neocavity.
  3. Perineal-scrotal reconstruction with fascial facing and cutaneous flaps

SUMMARY:
Type of study: Case series. Universe of study: Records of patients with Fournier syndrome treated using the 3-stage reconstructive technique assigned and treated at the Mexican Social Security Institute: Regional General Hospital No. 1 of Mérida, Yucatán, during the years 2021-2024.

Population under study: Patients diagnosed with Fournier syndrome.

DETAILED DESCRIPTION:
The first surgical stage consists of damage limitation and extension analysis. In the second surgical stage, it was necessary to wash and prepare the area to be remodeled with the joint creation of the testicular resting space delimited by the fascia of the adductor muscles of the proximal lower limb. Finally, in the third surgical stage, the wound is remodeled and addressed. The surgery was performed in patients with extensive involvement that could not be resolved with minor surgery.

The 3-stage reconstructive technique can be summarized as follows:

1. Analysis and limitation of the tissue injury. Bilateral testicular and spermatic cord dissection.
2. Formation of cutaneous flaps and bilateral inguinal neocavity.
3. Perineal-scrotal reconstruction with fascial facing and cutaneous flaps

ELIGIBILITY:
Inclusion Criteria:

- patients diagnosed with perineal necrotizing fasciitis (Fournier syndrome), at the General Hospital Zone No. 1, aged between 40-85 years, who have undergone surgery

Exclusion Criteria:

* Those who could not be followed up due to incomplete records. Those who did not complete the three procedures due to mortality associated with primary pathologies independent of necrotizing fasciitis.

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | From the diagnosis to the surgery and 30 day post op
  To determine the presence of mortality in patients with Fournier syndrome who underwent surgery using the 3-stage reconstructive technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Mexican Social Security Institute: Regional General Hospital No. 1, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
due to the reproducibility of the study

REFERENCES:
- [Background] Michael P, Peiris B, Ralph D, Johnson M, Lee WG. Genital Reconstruction following Fournier's Gangrene. Sex Med Rev. 2022 Oct 1;10(4):800-812. doi: 10.1016/j.sxmr.2022.05.002. PMID 37051973
- [Background] Lewis GD, Majeed M, Olang CA, Patel A, Gorantla VR, Davis N, Gluschitz S. Fournier's Gangrene Diagnosis and Treatment: A Systematic Review. Cureus. 2021 Oct 21;13(10):e18948. doi: 10.7759/cureus.18948. eCollection 2021 Oct. PMID 34815897
- [Background] Singh A, Ahmed K, Aydin A, Khan MS, Dasgupta P. Fournier's gangrene. A clinical review. Arch Ital Urol Androl. 2016 Oct 5;88(3):157-164. doi: 10.4081/aiua.2016.3.157. PMID 27711086